CLINICAL TRIAL: NCT04349501
Title: A Phase II Biomarker Study of Restriction Spectrum Imaging (RSI) MRI in Patients With High-Risk, Localized Prostate Cancer Who Will Receive Radiotherapy and Androgen Deprivation Therapy
Brief Title: Biomarker Monitoring of Prostate Cancer Patients With RSI MRI (ProsRSI)
Acronym: ProsRSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tyler Seibert, Assistant Professor, Radiation Medicine and Applied Sciences, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200266
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A logistic regression model of biochemical recurrence within 3 years will be fit, using maximum likelihood, on the change in RSI cellularity index from MRI #1 to MRI #2 and relevant covariates such as demographics. Continuous variables will be splined; only main effects will be considered. The cross-validated Area Under the Curve (AUC) for this model will be reported with a 95% bootstrap confidence interval using Efron's bias-corrected and accelerated (bca) method. If the lower bound on the 95% confidence interval of the Area Under the Curve (AUC) excludes 0.55, RSI cellularity index will be declared "viable" for identifying participants who will recur within the three-year post treatment. If declared "viable", a Cox model for predicting recurrence time will be fit, and the hazard ratios for RSI will be used to describe the adjusted associations supported by the data between RSI cellularity index and recurrence time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSI-MRI (Experimental): Participants will undergo RSI-MRI at three time points: before androgen deprivation therapy (ADT); after neoadjuvant ADT but before radiation therapy (RT); and after RT.
  Interventions: Other: Restriction Spectrum Imaging Magnetic Resonance Imaging

INTERVENTIONS:
Other: Restriction Spectrum Imaging Magnetic Resonance Imaging — RSI is a multicompartment model of diffusion MRI that uses data acquired at multiple b-values to distinguish varied diffusion speeds (restricted intracellular, hindered extracellular, and approximately free diffusion).
  Other Names: RSI-MRI

SUMMARY:
Adult male patients with high-risk, localized prostate cancer and planning to undergo radiation therapy (RT) with androgen deprivation therapy (ADT) will undergo an advanced Magnetic Resonance Imaging (MRI) examination called Restriction Spectrum Imaging (RSI-MRI) to evaluate whether RSI-MRI can predict treatment response.

DETAILED DESCRIPTION:
Participants will undergo RSI at three time points: before therapy (MRI #1), after neoadjuvant ADT (MRI #2), and after radiotherapy (MRI #3). Treatment response will be assessed primarily by absence of biochemical recurrence (PSA ≥2 ng/mL greater than nadir) within 3 years of completing radiotherapy. Change in RSI cellularity index from MRI #1 to MRI #2 will be evaluated for prediction of participants who will experience biochemical recurrence within 3 years, using area under the receiver operating characteristic curve. We hypothesize that RSI cellularity index will be an early biomarker for treatment effectiveness in prostate cancer treated with ADT and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥18 years, with histologically confirmed adenocarcinoma of the prostate
* High-risk prostate cancer (any of: PSA ≥20 ng/mL or cT3-T4 stage or Gleason score ≥8)
* Intended treatment and follow-up according to standard of care for prostate cancer
* Planning to undergo definitive radiotherapy with neoadjuvant and concurrent androgen deprivation therapy
* In good general health as evidenced by medical history and Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Prior radiotherapy to the pelvis
* Prior treatment for prostate cancer (cryotherapy, high frequency focused ultrasound, prostatectomy)
* Hip prosthesis
* Contraindication to MRI, per institutional requirements
* Technetium-99 bone scan showing no clear evidence of distant metastasis
* MRI or CT scan of the pelvis showing no clear evidence of bone or distant metastasis
* Another malignancy, unless in remission or unlikely to impact the patient's survival or ability to receive standard care for prostate cancer (e.g., cutaneous basal cell carcinoma)
* Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subjects undergoing treatment for Prostate Cancer
Enrollment: 100 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence (PSA 2 ng/mL greater than nadir) within 3 years of completing RT. | within 3 years of RT completion
  To evaluate the performance of the RSI cellularity index before and during therapy as a biomarker to identify participants who will experience biochemical recurrence within 3 years post-radiotherapy.

SECONDARY OUTCOMES:
PSA nadir within the 18 months after RT ≥0.5 ng/mL. | within 18 months of RT completion
  To evaluate the performance of the RSI cellularity index for identifying participants who will fail to reach a PSA nadir <0.5 ng/mL within 18 months of RT.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States